CLINICAL TRIAL: NCT00327158
Title: Using Transesophageal Echocardiography To Assess Fat Emboli As A Result Of Reaming In A Prospective Randomized Control Trial To Determine The Effectiveness Of Reaming In Diminishing Fat Emboli To The Lungs
Brief Title: A Prospective Study to Determine the Effectiveness of Reaming in Reducing Fat Emboli to the Lungs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Jeffrey Selby, UK Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0296-F1V
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Diaphyseal Femur Fracture
Keywords: Reaming; fracture; emboli
MeSH Terms: conditions — Fractures, Bone; Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transesophageal transducer — One time use of reamer during surgery
Procedure: echocardiography — takes photos of right atrium during the reaming processes

SUMMARY:
The purpose of the study is to see if there is a difference in the amount of fat droplets reaching the heart during surgery between the standard reamer currently used and a new reamer system which is expected to reduce the fat going into the blood, via an intraoperative echocardiography done through the food pipe.

DETAILED DESCRIPTION:
Reamed intramedullary nailing of diaphyseal femur fractures remains the standard of care for treatment of these fractures. Pressurization of the femoral canal during reaming leads to extra vasations of fat emboli into the systemic circulation, resulting in deposition of fat droplets in the pulmonary vasculature. This phenomenon has been well documented by use of Transesophageal Echocardiography. A novel reaming system has recently become available that may limit this phenomenon. The new reamer system incorporates irrigation and aspiration during reaming, theoretically minimizing pressurization and fat emboli. Additionally, this reamer system allows for one pass reaming as compared to the current system which requires multiple reaming passes.

The objective of this study is to determine effectiveness of reaming in diminishing fat emboli to the lungs as evidenced by decreased numbers of large fat droplets entering the right heart as measured by transesophageal echocardiography during the reaming process. This will determine if there is a benefit to aspiration during reaming as would be expected.

During the reaming process a transesophageal echo cardiogram will be performed to analyze the presence or absence of emboli and the mean regarding the total time that each of the embolic grades is present during each of the intervals across the patient groups

ELIGIBILITY:
Inclusion Criteria:

* diaphyseal femur fractures undergoing reamed intramedullary nailing
* male or female
* 18 years of age or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Presence of Emboli | Immediately following surgery

CONTACTS AND LOCATIONS:
Overall Officials: William Rosenblum, MD, Principal Investigator — University of Kentucky, Department of Orthopaedic Surgery; Jeffrey Selby, MD, Principal Investigator — University of Kentucky Department of Orthopaedic Surgery
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States